CLINICAL TRIAL: NCT06104475
Title: Diagnostic Performance of Chest Computed Tomography Scan in Patients Aged 65 and Over Presenting to Emergency Room With Acute Dyspnea
Acronym: CT-Dys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP220845
Record Dates: First submitted 2023-10-20; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Dyspnea
Keywords: Dyspnea; ED; Chest CT-scan
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT scan intervention (Experimental)
  Interventions: Other: CT scan

INTERVENTIONS:
Other: CT scan — A CT scan will be requested for every patient in addition to the chest X-ray

SUMMARY:
In acute dyspnea, the use of chest radiography is frequent and not very contributive, especially in the elderly patients.

However, early diagnosis of the cause of dyspnea in the ED is associated with a better prognosis, in particular for the identification of an infectious or cardiac origin.

Chest CT has already shown better diagnostic performances than conventional radiography in several pathologies such as low respiratory infection, and the development of so-called "low dose" scans allows to limit the irradiation during this examination.

The investigators aim to conduct a diagnostic study comparing non-injected chest CT-scan and conventional chest radiography in patients older than 65 presenting in the ED with acute dyspnea to assess whether CT-scan improves diagnosis.

DETAILED DESCRIPTION:
Patients of 65 years and older presenting to the emergency department with acute dyspnea and for whom a chest radiography is mandatory will be screened for inclusion. If the inclusion criteria are met and in the absence of non-inclusion criteria, free and informed oral consent will be sought.

Once the patient is included, management by the emergency physician will be routine.

A non-injected chest CT scan will be requested to the emergency radiology department in addition to the chest radiography. As a result, an X-ray and then a CT scan will be performed in each patient.

3 diagnoses will be collected:

1. By the emergency physician in charge of the patient, after the chest X-ray and before the CT scan (DiagU1)
2. By the emergency physician in charge of the patient, after the results of the scan (DiagU2)
3. By an adjudication committee after review of the medical file (DiagExpert) A comparison will be made between the 3 diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 65 years
* Acute dyspnea (< 1 week)
* Prescription of a chest x-ray
* Oral free and informed consent of the patient after information and delivery of the information note
* Patient affiliated to a social security system

Exclusion Criteria:

* Inability to lie down
* Chest imaging done within the last 7 days
* Indication to perform a thoracic scan
* Patient under guardianship or curatorship
* Patient deprived of liberty, pregnant woman
* Participation in other interventional research

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Improved diagnosis | 28 days after inclusion
  Proportion of patients with "bad diagnosis" before scanning and "good diagnosis" after scanning (according to adjudication committee)

SECONDARY OUTCOMES:
Discordant diagnosis | 28 days after inclusion
  Proportion of patients with discordant pre- and post-scan diagnoses
Improvement in diagnostic certainty | 28 days after inclusion
  Difference in "Diagnostic certainty" in percentage by self-assessment before and after scan
Scans performed | baseline (Day 0)
  Proportion of patients for whom the scan was actually performed

CONTACTS AND LOCATIONS:
Overall Officials: Yonathan FREUND, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Emergency department Hospital Pitié-Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No